CLINICAL TRIAL: NCT05433311
Title: The Effect of Exercise Program on Perception of Exercise and Fear of Movement in Nonspecific Low Back Pain
Brief Title: The Effect of Exercise on Motion Perception and Fear in Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Mine ARGALI DENIZ, PhD, Clinical Physiotherapist, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 72867572-050.01.04-95550
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Low Back Pain
Keywords: nonspesific low back pain; flexibility; kinesiphobia; pain
MeSH Terms: conditions — Low Back Pain; Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Patients included in the treatment group had 15 sessions. Neutral position training, transversus abdominis/multifidius/abdominal/back extensors strengthening exercise, bridge exercise, cat-camel exercise, lumbal extensor/hamstring/gastrosoleus/latissimus dorsi/gluteal stretching exercises will be done face-to-face with a physiotherapist. At the end of the 15 sessions of face-to-face training the patients will be perform the same exercises at home for 15 days. The patients will not given any exercises in the control group. Measurements and evaluations of the patients in the both groups will be made three that pre-treatment, post-treatment, 15 days after the end of treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercises (Active Comparator): Neutral position training, transversus abdominis/multifidius/abdominal/back extensors strengthening exercise, bridge exercise, cat-camel exercise, lumbal extensor/hamstring/gastrosoleus/latissimus dorsi/gluteal stretching exercises
  Interventions: Other: Exercises
- Routine (No Intervention): Only routine treatment

INTERVENTIONS:
Other: Exercises — Neutral position training, transversus abdominis/multifidius/abdominal/back extensors strengthening exercise, bridge exercise, cat-camel exercise, lumbal extensor/hamstring/gastrosoleus/latissimus dorsi/gluteal stretching exercises
  Arms: Exercises

SUMMARY:
Nonspesific low back pain (NLBP), which negatively affects functionality, activity participation, and financial situation, is now one of the leading causes of disability in the world. In NLBP, pain causes kinesiophobia known as fear of movement and limitation of activity. Contrary to what is known, this cycle aggravates pain. With this result, it is suggested that the exercise to be done will improve the perception of benefit in the person and eliminate the fear of movement, and that it will cure the disease. In this context, the aim of the study is to examine the effect of exercise on the perception of exercise and fear of movement in patients with NLBP.

DETAILED DESCRIPTION:
The study will be composed of volunteers, non-specific low back pain individuals who meet the inclusion criteria. First of all, the demographic and clinical characteristics of the patients will be questioned with the evaluation form. The personal information of the patients (gender, height, weight, smoking, etc.) and clinical status (pain type, pain intensity, trunk flexibility measurements) will be recorded by the physiotherapist in the evaluation form. In addition to these measurements, the state of fear of physical movement and activity will be evaluated with the Tampa Kinesiophobia Scale.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily accepting the study
* Having nonspecific low back pain for 3 months or longer
* Not having had spinal surgery in the last 6 months
* Not having an orthopedic or neurological disability that would prevent them from doing their exercises
* Patients who regularly continue their exercises without interrupting

Exclusion Criteria:

* Patients with non-specific low back pain who do not meet the inclusion criteria and want to drop out of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-06 (Actual); Primary Completion 2022-09-20 (Estimated); Study Completion 2022-12-25 (Estimated)

PRIMARY OUTCOMES:
Exercise Benefit/Barrier Scale | Change in participate in life ine one month
  This scale is a 4 scores Likert-type. Scale consisting 43 questions. A high score means exercise perception. When Benefit Scale is evaluated on its own, how high the total score of 29 items is it means that exercise perception is beneficial in high level. In Barrier Scale which consists 14 items, the higher obtained total score is, higher the barrier level perceived against exercise is.

SECONDARY OUTCOMES:
Tampa Scale of Kinesiophobia | Change in participate in life ine one month
  Tampa Scale of Kinesiophobia is a checklist of 17 questions. 4-point Likert scale on the scale rating (1= strongly disagree, 4= I totally agree). Person between 17-68 total gets a score. The score of the person on the scale high, kinesiophobia is also high. shows. Total score in studies use is recommended.

CONTACTS AND LOCATIONS:
Overall Officials: Mine ARGALI DENIZ, PT, PhD, Study Director — Suleyman Demirel University Education and Training Hospital
Locations (1):
- Mine ARGALI DENIZ, Isparta, Turkey (Türkiye)